CLINICAL TRIAL: NCT03804281
Title: Clinical Evaluation of Gingival Margin Stability Following Conventional Versus Microsurgical Techniques of Esthetic Crown Lengthening
Brief Title: Clinical Evaluation of Conventional Versus Microsurgical Techniques of Esthetic Crown Lengthening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed elshafie mohamed tawfiq hassan, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dentaris192018
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Gummy Smile
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): esthetic crown lengthening with microsurgical approach
  Interventions: Procedure: Test group
- Control group (Active Comparator): esthetic crown lengthening with conventional approach.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Test group — The surgery will be done with the use of 4x magnification loop, the knives are micro blades and micro-sutures 7//0 used with the microsurgical instruments kit
  Arms: Test group
Procedure: Control group — esthetic crown lengthening with conventional approach with an internal bevel incision, following CEJ anatomy, this will be followed by an intra-sulcular incision, removal of the strip of outlined marginal gingiva and elevation of a mucoperiosteal ﬂap to the level of the alveolar bone crest.
  Arms: Control group

SUMMARY:
the study compare gingival margin stability following conventional approach versus microsurgical approach of esthetic crown lengthening in management of patients with short clinical crowns in the upper anterior region.In management of patients with short clinical crowns in the upper anterior region, there is no difference in gingival margin stability between conventional and microsurgical approaches of esthetic crown lengthening.

ELIGIBILITY:
Inclusion Criteria:

* Patients with healthy systemic condition.
* Adult patients ˃ 18 years old.
* The presence of the six upper anterior teeth.
* Absence of sites with attachment loss and probing depth (PD) >3 mm
* Keratinized gingiva of at least 2mm width.
* Compliance with good oral hygiene.
* Patients accepts 6-months follow-up period (cooperative patients).
* Patients provides an informed consent

Exclusion Criteria:

* Gummy smile with normal tooth proportions
* Presence of prosthetic crowns
* Extensive restorations
* Extensive incisal edge attrition.
* Misalignment on maxillary anterior teeth.
* Smokers ˃ 10 cigarettes / day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Mid-buccal gingival margin level | 6 months
  periodontal probe with William's graduation will be used to measure the distance from the CEJ to the gingival margin at the mid-buccal surface

SECONDARY OUTCOMES:
Pink Esthetic Score (PES) | 6 months
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable shall be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. The mesial and distal papilla will be evaluated for completeness, incompleteness or absence
Post-Surgical swelling | 7days
  will be evaluated post-surgically with Verbal Rating Scale with words ranging from (absent-slight-moderate-intense) Absent (no swelling), Slight (intraoral swelling at the operated area), Moderate (moderate intraoral swelling at the operated area) and Intense (intensive extra oral swelling extending beyond the operated area).
Post-Surgical Patient Satisfaction: 3-item questionnaire | 6 months
  A 3-item questionnaire is asked and the patients shall use a 7-point answer scale

IPD SHARING:
Plan to Share IPD: Undecided